CLINICAL TRIAL: NCT00859040
Title: Phase II Study of Monthly SOM230C for Recurrent or Progressive Meningioma
Brief Title: Monthly SOM230C for Recurrent or Progressive Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Memorial Sloan Kettering Cancer Center (Other); Wake Forest University Health Sciences (Other); Duke University (Other); Cedars-Sinai Medical Center (Other); Northwestern University (Other); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Directory, Center for Neuro-Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-266; CSOM230CUS09T
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Meningioma
Keywords: recurrent intracranial meningioma(s); progressive intracranial meningioma(s)
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOM230C (Experimental): Monthly SOM230C (pasireotide LAR) - 60 mg intramuscularly (Single-Arm Trial)
  Interventions: Drug: SOM230C

INTERVENTIONS:
Drug: SOM230C — Injection in the buttocks every 28 days
  Other Names: pasireotide LAR

SUMMARY:
The purpose of this research study is to evaluate the effectiveness and safety of SOM230C in treating recurrent meningiomas. SOM230C is a newly discovered drug that may stop meningioma cells from growing abnormally. This drug has been used in treatment of other tumors, and information from those other research studies suggests that SOM230C may help to stop the growth of meningiomas.

DETAILED DESCRIPTION:
* To enroll in the study, a sample of the participant's tumor tissue, stored from an earlier study, must be sent to a lab at the Dana-Farber/Harvard Cancer Center for diagnosis and special testing.
* Prior to starting the study medication, participants will undergo a Octreotide scan. This is a special type of scan used to obtain information about certain tumors.
* Participants will receive the study medication, SOM230C, via an injection into the buttocks every 28 days. Therefore, each treatment cycle lasts 28 days.
* The following tests and procedures will be done prior to the first, second and third treatment cycles, and every three treatment cycles thereafter: Complete physical examination including neurological exam; vital signs; current medication and symptom review; blood samples and a pregnancy test (for women of child-bearing potential).
* About 2/3 through the first treatment cycle (around day 22), participants will visit the research doctor for a complete physical examination including a neurological exam and blood work.
* Participants will have ECGs done prior to their first treatment cycle, about 2/3 through the first and third treatment cycles (around day 22), prior to their sixth treatment cycle, and every three treatment cycles thereafter.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Radiographically measurable disease on contrast-enhanced MRI or CT images
* Karnofsky Performance status of 60 or greater
* Life expectancy of at least 3 months
* Histologically confirmed diagnosis of recurrent or progressive intracranial meningioma(s). This includes benign, atypical, or malignant meningioma; patients with neurofibromatosis type 1 or 2 may participate. Participants without histological confirmation but a classic radiographic picture of meningioma may also enroll. Patients with neurofibromatosis type 2 and a classic radiographic picture of meningioma may also enroll without histological confirmation
* At least ten unstained standard (4-5 micron) paraffin slides for immunohistochemistry. Participants who have not had a surgical procedure are exempt from this requirement
* Unequivocal evidence for tumor progression by MRI (or CT scan if MRI is contraindicated)
* MRI or CT must be performed within 14 days of registration
* Patients with malignant meningiomas who require corticosteroids must be on a stable dose for at least 5 days prior to baseline imaging.
* For patients who have been treated with external beam radiation, interstitial brachytherapy, or radiosurgery, an interval of 4 or more weeks must have elapses from the completion of radiation therapy to study drug administration, and there must be evidence of tumor progression.
* There is no limit on the number of prior therapies

Exclusion Criteria:

* Any cytotoxic chemotherapy, radiation, immunotherapy, or experimental therapy within 4 weeks prior to study drug administration
* Prior therapy with somatostatin, andy somatostatin analogue, or any other hormonal treatment prescribed for the purpose of treating meningioma
* Major surgery within 4 weeks prior to study drug administration
* Malabsorption syndrome, short bowel or chologenic diarrhea not controlled by specific therapeutic means
* Poorly controlled diabetes mellitus
* Symptomatic cholelithiasis
* Congestive heart failure, unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment
* QTc > 450 msec
* Risk factors for Torsades de Pointes such as hypokalemia (< 3.5 mmol/L) not corrected by treatment, hypomagnesemia (< 0.7 mmol/L or < 1.6 mg/dL) not corrected by treatment, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
* Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Concomitant medication(s) known to increase the QT interval within 4 weeks prior to study drug administration
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis with serum bilirubin > 2x ULN, serum albumin < 0.67 LLN, or ALT or AST more than 2 x ULN
* Any other primary malignancy within the past 3 years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)
* Active or suspected acute or chronic, uncontrolled infection or any history of immunocompromise, including any positive HIV test result
* Abnormal coagulation studies (PT or PTT elevated by 30% above normal limits)
* Use of anticoagulant medications (not including anti-platelet medications)
* Lab values as specified in the protocol
* Any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator
* Pregnancy or lactation, or failure to practice a medically acceptable method of birth control
* History of alcohol or drug abuse in the 6 month period before study enrollment
* Participation in any clinical investigation with an investigational drug within 1 month prior to study drug administration
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR os s.c. formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Preston Robert Tisch Brain Tumor Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Atypical/Malignant Meningiomas: participants with atypical meningiomas (WHO grade 2) or malignant meningiomas (WHO grade 3): patients receive SOM230C (pasireotide LAR) 60 mg intramuscular injections in the buttocks every 28 days
- Participants With Benign Meningiomas: participants with benign meningiomas (WHO grade 1) or meningiomas with undetermined histology: patients receive SOM230C (pasireotide LAR) 60 mg intramuscular injections in the buttocks every 28 days
Period: Overall Study
Arm/Group | Participants With Atypical/Malignant Meningiomas | Participants With Benign Meningiomas
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Atypical/Malignant Meningiomas | Participants With Benign Meningiomas | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 74] | 52 [36 to 81] | 54 [36 to 81]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White, Non-Hispanic | 14 | 15 | 29
  Black or African American, Non-Hispanic | 3 | 0 | 3
  Hispanic or Latino (Unknown Race) | 1 | 0 | 1
  White (Unknown Ethnicity) | 0 | 1 | 1
KPS scores [Median (Full Range); unit: percent] — 100% = Normal; 90% = Normal activity, minor signs/symptoms; 80% = Normal activity w/ effort, some signs/symptoms; 70% = Cares for self, unable to do normal activity/active work; 60% = Requires occasional assistance, but cares for most personal needs; 50% = Requires considerable assistance/frequent medical care; 40% = Disabled, requires special care & assistance; 30% = Severely disabled, hospital admission is indicated but death not imminent; 20% = Very sick, hospitalization necessary, active supportive treatment necessary; 10% = Moribund, fatal processes progressing rapidly; 0% = Dead.
  percent | 80 [60 to 100] | 90 [70 to 100] | 85 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival
Description: Progression is defined using Modified Macdonald Criteria , using a >/= 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR clear clinical worsening or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Participants With Atypical/Malignant Meningiomas | Participants With Benign Meningiomas
Number analyzed (Participants) | 18 | 16
percentage of patients | 11 | 44

2. Secondary Outcome: Response Rate
Description: Number of participants to experience complete or partial response on study treatment.
  For response per Modified Macdonald Criteria, all measurable and evaluable lesions and sites must be assessed using the same techniques as baseline.
  1. Complete Response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients must be on no steroids.
  2. Partial Response (PR): Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. The steroid dose at the time of the scan evaluation should be no greater than the maximum dose used in the first 8 weeks from initiation of therapy.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Participants With Atypical/Malignant Meningiomas | Participants With Benign Meningiomas
Number analyzed (Participants) | 18 | 16
participants | 0 | 0

3. Secondary Outcome: Treatment-related Events
Description: All Grade 3-4-5 adverse events with a treatment attribution of probable, possible or definite based on CTCAE (v3.0) as reported on case report forms
Time Frame: 5 years
Measure: Number; unit: events
Arm/Group | SOM230C
Number analyzed (Participants) | 34
events
  Amylase | 1
  Fatigue | 2
  Hyperglycemia | 8
  Hypoglycemia | 1
  Hypokalemia | 1
  Lipase | 3

4. Secondary Outcome: Median Progression-Free Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Participants With Atypical/Malignant Meningiomas | Participants With Benign Meningiomas
Number analyzed (Participants) | 18 | 16
weeks | 15 [8 to 20] | 26 [12 to 43]

5. Secondary Outcome: Median Time to Progression
Description: Per protocol, the study's secondary objectives are to be evaluated "for the estimate of median ... PFS ... at time of interest." At this time, all study participants have been followed for progression for a minimum of 34 months (final patient to accrue to study was registered to trial on 06/14/2011), and study manuscript is currently being written-up with this information.
Time Frame: 34 months
Population: Time to progression only reported for the 32 patients who have progressed (either on treatment or in follow-up).
  [NOTE: The other 2 patients who were treated on study each remain progression-free after > 1000 days.]
Measure: Median (Full Range); unit: days
Arm/Group | SOM230C
Number analyzed (Participants) | 32
days | 124 [43 to 645]

6. Secondary Outcome: Overall Survival
Description: Percentage of participants alive 34 months after initiating study treatment. Median Overall Survival has not yet been reached for one study group; therefore, we are reporting Overall Survival rates by the end of the study time frame.
Time Frame: 34 months
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Atypical/Malignant Meningiomas | Participants With Benign Meningiomas
Number analyzed (Participants) | 18 | 16
percentage of participants | 45 | 73

ADVERSE EVENTS:
Arm/Group | SOM230C
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230C (N=34)
somnolence (Nervous system disorders) | 1 (1) — grade 3 somnolence with vomiting and left-sided weakness resulting in hospitalization (unlikely related to & unexpected with SOM230C)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1) — grade 4 hypoglycemia (w/ hospitalization), with anemia (grade 3 hemoglobin); unrelated to and unexpected with SOM230C.
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — grade 4 hyperglycemia (w/ hospitalization); definitely related to and expected with SOM230C.
subdural hematoma (Vascular disorders) | 1 (1) — grade 4 subdural hematoma (w/ hospitalization); unrelated to and unexpected with SOM230C
secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — grade 3 secondary malignancy (squamous cell carcinoma); unrelated to and unexpected with SOM230C.
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Gr 3 lower extremity weakness/decline (w/ hosp); unrelated & unexpected.
extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 3 lower extremity (gait/walking) complications (w/ hospitalization); unrelated to and unexpected with SOM230C.
sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) — grade 3 hyponatremia w/ hallucinations (w/ hospitalization); unrelated to and unexpected with SOM230C.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOM230C (N=34)
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 7
Leukocytes (Blood and lymphatic system disorders) | 3
Neutrophils (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 4
QTc interval (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 3
Constitutional - Other (General disorders) | 3
Fatigue (General disorders) | 16
Insomnia (General disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Skin - Other (Skin and subcutaneous tissue disorders) | 4
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 15
Dysphagia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 8
GI - Other (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Taste DIsturbance (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Infection Gr0-2 neut- upper airway (Infections and infestations) | 2
Infection Gr0-2 neut- urinary tract (Infections and infestations) | 2
Infection - Other (Infections and infestations) | 2
Alkaline phosphatase (Investigations) | 3
ALT - SGPT (Investigations) | 3
Amylase (Investigations) | 5
AST - SGOT (Investigations) | 2
Creatinine (Investigations) | 2
GGT (Investigations) | 3
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 8
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 16
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 4
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3
Lipase (Investigations) | 4
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 4
Extremity-lower (gait/walking) (General disorders) | 6
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic right-side muscle weak (Musculoskeletal and connective tissue disorders) | 2
Mood Alteration: Anxiety (Psychiatric disorders) | 3
Ataxia (Nervous system disorders) | 7
Cognitive disturbance (Nervous system disorders) | 3
Confusion (Psychiatric disorders) | 3
Mood Alteration: Depression (Psychiatric disorders) | 3
Dizziness (Nervous system disorders) | 3
Memory Impairment (Nervous system disorders) | 5
Neurologic - Other (Nervous system disorders) | 5
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 5
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 7
Speech Impairment (Nervous system disorders) | 4
Ocular - Other (Eye disorders) | 3
Pain - Abdomen NOS (Gastrointestinal disorders) | 4
Pain - Back (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity/Limb (Musculoskeletal and connective tissue disorders) | 4
Pain - face (General disorders) | 2
Pain - head/headache (Nervous system disorders) | 21
Pain - oral cavity (Gastrointestinal disorders) | 2
Pain - other (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2
Incontinence, urinary (Renal and urinary disorders) | 3
Renal/GU - Other (Renal and urinary disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days